CLINICAL TRIAL: NCT03400137
Title: Effects of Elevated Intraocular Pressure on the Lamina Cribrosa
Brief Title: IOP Elevation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-01027; R01EY013178 (NIH)
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Healthy Volunteers (Active Comparator): No family history (first degree relative) of glaucoma.
  Interventions: Diagnostic Test: Increasing of intraocular pressure (IC)
- Glaucoma suspects (Active Comparator): oEither IOP between 25 to 30 mmHg with central corneal thickness < 550µm, or a difference ≥ 0.2 in cup to disc ratio between eyes.
  Interventions: Diagnostic Test: Increasing of intraocular pressure (IC)
- Glaucoma (Active Comparator): Rim thinning, notching, undermining (excavation) or diffuse or localized RNFL defects that are characteristic of glaucoma.
  Interventions: Diagnostic Test: Increasing of intraocular pressure (IC)

INTERVENTIONS:
Diagnostic Test: Increasing of intraocular pressure (IC) — intraocular pressure will be increased using an ophthalmodynanometer

SUMMARY:
The purpose of this study is to improve understanding of the pathophysiologic process that leads to the development of glaucamotous damage. The mechanism by which vision loss in glaucoma occurs is still unknown, but it is clear that increased intraocular pressure (IOP) is a major risk factor. It is also thought that the LC is a site of primary damage during pathogenesis of the disease. This prospective study with determine the in-vivo mechanical response to IOP modulation at the level of the ONH and LC.

DETAILED DESCRIPTION:
The present study will briefly increase the pressure in eyes of living subjects and examine the effect of elevated intraocular pressure on optic nerve topography and position during pressure elevation using optical coherence tomography imaging of the posterior eye. Outcome measures will include measurements in microns based on these images quantifying the deformation of the lamina cribrosa.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

* No family history (first degree relative) of glaucoma.
* No history of IOP >22 mmHg.
* Normal appearing optic discs and RNFL on dilated fundus examination.
* Normal Swedish interactive thresholding algorithm (SITA) standard perimetry tests as defined by glaucoma hemifield test (GHT) within normal limits.

Glaucoma suspects

* Normal visual field as defined above.
* Either IOP between 25 to 30 mmHg with central corneal thickness < 550µm, or a difference ≥ 0.2 in cup to disc ratio between eyes.

Glaucoma

* Glaucomatous ONH abnormality: rim thinning, notching, undermining (excavation) or diffuse or localized RNFL defects that are characteristic of glaucoma.
* Two consecutive abnormal SITA standard perimetry tests with GHT outside normal limits.

Exclusion Criteria:

* Media opacity (e.g. lens, vitreous, cornea).
* Strabismus, nystagmus or a condition that would prevent fixation.
* Diabetes with evidence of retinopathy.
* Previous intraocular surgery or ocular trauma (with the exception of laser procedures and subjects that have undergone uneventful cataract surgery more than 6 months from enrollment date).
* Neurological and non-glaucomatous causes for visual field damage.
* Any intraocular non-glaucomatous ocular disorders.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2024-05-08 (Estimated); Study Completion 2024-05-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of the deformation of the lamina cribrosa in healthy eye in response to increasing intraocular pressure. | 10 Minutes
  OCT scanning will be obtained at baseline and with increased IOP. The IOP elevation will last no longer than two minutes, during which scans will be acquired by the imaging device.
Assessment of the deformation of the lamina cribrosa in glaucoma suspect, in response to increasing intraocular pressure. | 10 Minutes
  OCT scanning will be obtained at baseline and with increased IOP. The IOP elevation will last no longer than two minutes, during which scans will be acquired by the imaging device.
Assessment of the deformation of the lamina cribrosa in glaucomatous eyes in response to increasing intraocular pressure. | 10 Minutes
  OCT scanning will be obtained at baseline and with increased IOP. The IOP elevation will last no longer than two minutes, during which scans will be acquired by the imaging device.

CONTACTS AND LOCATIONS:
Overall Officials: Gadi Wollstein, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States